CLINICAL TRIAL: NCT04405089
Title: Role of Transcranial Direct Current Stimulation to Decrease Impulsivity and Compulsivity in Individuals With Obesity
Brief Title: tDCS for Impulsivity and Compulsivity in Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Center for Veterans Research and Education (Other)
Responsible Party: Principal Investigator, Shalamar Sibley, MD, MPH, Associate Professor of Medicine, University of Minnesota; Minneapolis VAMC Staff Physician, Minneapolis Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4740A
Record Dates: First submitted 2020-05-17; First posted 2020-05-28 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Impulsivity; Compulsive Overeating; Obesity
Keywords: Impulsive Behavior; Behavior Control; Appetitive Behavior; Health Risk Behaviors; Compulsive Behavior
MeSH Terms: conditions — Impulsive Behavior; Obesity; Appetitive Behavior; Health Risk Behaviors; Compulsive Behavior | interventions — Transcranial Direct Current Stimulation; Cognitive Training

STUDY DESIGN:
Intervention Model Description: The study is not a disease treatment study. It involves of an Non-Significant Risk (NSR) device coupled with a set of computerized cognitive tasks in a small group of participants with primary outcome of change in an NIH Examiner domain (Flanker).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active tDCS with cognitive training (Experimental): Participants will receive 5 sessions of cognitive training concurrent with transcranial direct current stimulation (anode over right frontal cortex, cathode over left frontal cortex; 2 mAmps for 26 minutes).
  Interventions: Device: Device: Active Transcranial Direct Current Stimulation (tDCS) coupled with cognitive training
- Sham tDCS with cognitive training (Sham Comparator): Participants will receive 5 sessions of cognitive training concurrent with sham tDCS. For sham tDCS, electrodes are placed at the same locations as for active tDCS, but current is ramped up for the initial 30 secs, then immediately ramped back down. This method mimics the initial physical sensation of stimulation, but there is no active current for the remainder of the session.
  Interventions: Device: Device: Sham Transcranial Direct Current Stimulation (tDCS) coupled with cognitive training

INTERVENTIONS:
Device: Device: Active Transcranial Direct Current Stimulation (tDCS) coupled with cognitive training — Cognitive training concurrent with 2 milliamperes (mAmps) of anodal stimulation applied to the right prefrontal cortex for total of 26 minutes.
  Arms: Active tDCS with cognitive training
Device: Device: Sham Transcranial Direct Current Stimulation (tDCS) coupled with cognitive training — Cognitive training concurrent with sham tDCS (30 secs ramp up/ramp down of current at beginning of session).
  Arms: Sham tDCS with cognitive training

SUMMARY:
Even when they know it can improve health, many individuals with loss of control eating struggle when they are trying to make and sustain new health habits for weight loss and maintenance of weight loss. Impulsivity, characterized by lack of foresight and planning and excessive risk taking, and compulsivity, characterized by inability to break old habitual behaviors, may play a role in refractory obesity. The primary objective of this pilot study is to investigate the effect of a novel neuroplasticity based intervention, cognitive training coupled with transcranial direct current stimulation (tDCS), on measures of impulsivity and compulsivity in individuals with obesity.

DETAILED DESCRIPTION:
Impulsivity and compulsivity are two psychological factors which contribute to addictive behaviors. Impulsivity is characterized by lack of foresight and planning, and excessive risk taking. Impulsivity is a characteristic of poor executive functioning, and reflects deficits in goal-oriented behavior and self-regulation. Compulsivity is characterized by inability to break old habits. Both of these traits may play a role in refractory obesity. Transcranial direct current stimulation (tDCS) coupled with cognitive training may strengthen key circuitry involved in impulse control within the prefrontal cortex. tDCS coupled with cognitive training has the potential to reduce impulsivity and compulsivity in individuals with obesity, with the potential for therapeutic application as a non-pharmacologic approach to management of food-related eating behaviors which may impact weight.

For this double-blind, randomized, placebo (sham) controlled study pilot study the investigators aim to recruit and complete studies in approximately 20 individuals, randomly assigned to receive either active or sham tDCS, both coupled with computerized cognitive training tasks, for five days. Additionally, participants will attend follow up visits at approximately 2, and 4 months after the course of intervention visits is completed. Testing pre- and post-intervention will include the Binge Eating Scale (BES), Patient Health Questionnaire 9 (PHQ-9) Depression Screen, and 4 domains of the NIH Examiner Battery. Weight will be tracked throughout the study. The Minnesota Blast Exposure Screening Tool (MN-BEST) is also conducted at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Obese (BMI>30)
* Adults ages 18 years or older receiving care through the Minneapolis VA Healthcare System
* Able to understand English, self-consent and follow study-related procedures
* Willing to use a reliable form of birth control if they are of females of child-bearing potential.

Exclusion Criteria:

* History of any of the following issues: seizures, severe or moderate head injury, head surgery, significant neurological disorder(significance based on Principal Investigator's judgment), frequent severe headaches
* History of scalp conditions such as eczema or seborrheic dermatitis
* Metal in head (other than in mouth) including shrapnel/surgical clips/welding fragments
* Implanted medical devices (including pumps and cardiac pacemakers)
* Pregnancy
* Active substance abuse
* Psychological or medical disorders requiring inpatient treatment
* Presence of a known metabolic or hormonal disorder (such as Cushing's) which affects weight/appetite. (History of hypothyroidism is acceptable if subject is on treatment with normal thyroid stimulating hormone (TSH) and free thyroxine (FT4) on most recent check within the last 3 months and has been on stable dosage of l-thyroxine for at least 3 months, taking it as prescribed.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shalamar Sibley, MD, MPH, Principal Investigator — Minneapolis VAMC, University of Minnesota
Locations (1):
- Minneapolis VA Medical Center, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment/follow up completed with final participant's final visit (visit 8) on 6/26/20.
Groups:
- Active tDCS With Cognitive Training: Participants received 5 sessions of cognitive training concurrent with transcranial direct current stimulation (anode over right frontal cortex, cathode over left frontal cortex; 2 milliamperes (mAmps) for 26 minutes).
  Device: Active Transcranial Direct Current Stimulation (tDCS) coupled with cognitive training: Cognitive training concurrent with 2 mAmps of anodal stimulation applied to the right prefrontal cortex for total of 26 minutes.
- Sham tDCS With Cognitive Training: Participants received 5 sessions of cognitive training concurrent with sham tDCS. For sham tDCS, electrodes are placed at the same locations as for active tDCS, but current is ramped up for the initial 30 secs, then immediately ramped back down. This method mimics the initial physical sensation of stimulation, but there is no active current for the remainder of the session.
  Device: Sham Transcranial Direct Current Stimulation (tDCS) coupled with cognitive training: Cognitive training concurrent with sham tDCS (30 secs ramp up/ramp down of current at beginning of session).
Period: Overall Study
Arm/Group | Active tDCS With Cognitive Training | Sham tDCS With Cognitive Training
Started | 15 | 16
Completed | 8 | 9
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Population: Two participants who were randomized to a group but did not start study intervention were included in this table.
Groups:
- Active tDCS With Cognitive Training: Participants receive 5 sessions of cognitive training concurrent with transcranial direct current stimulation (anode over right frontal cortex, cathode over left frontal cortex; 2 mAmps for 26 minutes).
  Device: Active Transcranial Direct Current Stimulation (tDCS) coupled with cognitive training: Cognitive training concurrent with 2 mAmps of anodal stimulation applied to the right prefrontal cortex for total of 26 minutes.
- Sham tDCS With Cognitive Training: Participants receive 5 sessions of cognitive training concurrent with sham tDCS. For sham tDCS, electrodes are placed at the same locations as for active tDCS, but current is ramped up for the initial 30 secs, then immediately ramped back down. This method mimics the initial physical sensation of stimulation, but there is no active current for the remainder of the session.
  Device: Sham Transcranial Direct Current Stimulation (tDCS) coupled with cognitive training: Cognitive training concurrent with sham tDCS (30 secs ramp up/ramp down of current at beginning of session).
- Total: Total of all reporting groups
Arm/Group | Active tDCS With Cognitive Training | Sham tDCS With Cognitive Training | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 20
  >=65 years | 4 | 7 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 9 | 12 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 12 | 13 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Flanker Task Reaction Time [Mean (Standard Deviation); unit: seconds] — In the Flanker Task, a participant is instructed to press a key in response to viewing a stimulus presented on-screen. The Reaction Time, or the amount of time in seconds between presentation of the stimulus and the response, is measured.
  seconds | 0.86 (0.17) | 0.89 (0.21) | 0.88 (0.19)
Set Shifting Task Score [Mean (Standard Deviation); unit: score on a scale] — Description: The Set Shift Task Score is an ultimate composite score that is a summary score of reaction time and accuracy sub-scales. Scale range: Minimum 0, Maximum 10. Higher values represent a better outcome.
  score on a scale | 7.73 (0.93) | 7.65 (0.76) | 7.69 (0.83)
Unstructured Task Score [Mean (Standard Deviation); unit: score on a scale] — The Unstructured Task Score is the total sum of points awarded for completed puzzle items. Scale range: Minimum 0, Maximum 1469. Higher values represent a better outcome. The total score is a sum of scores for 3 individual trials.
  score on a scale | 336.07 (66.11) | 328.44 (91.11) | 332 (79.17)
Dot Counting Task Score [Mean (Standard Deviation); unit: score on a scale] — The Dot Count Task Score is the total sum of points awarded for dots a participant counts on the screen. Scale range: Minimum 0, Maximum 27. Higher values represent a better outcome. The total score is a sum of scores for 27 individual trials.
  score on a scale | 14.64 (4.41) | 15.25 (4.23) | 14.97 (4.25)
Weight [Mean (Standard Deviation); unit: pounds] | 260.76 (59.33) | 251.95 (44.46) | 256.06 (51.19)

OUTCOME MEASURES:

1. Primary Outcome: Change in NIH Examiner Flanker Task Reaction Time
Description: Differences in change in Flanker Task reaction time (score at final follow-up visit minus score at baseline) between active tDCS-cognitive training and sham-cognitive training groups.
  NIH Flanker absolute value range: 0 to 5 seconds. Higher values represent a better outcome.
  In the Flanker Task, a participant is instructed to press a key in response to viewing a stimulus presented on-screen. The Reaction Time, or the amount of time in seconds between presentation of the stimulus and the response, is measured.
Time Frame: Change between baseline and 4 months post-stimulation (timepoint 8/final visit)
Population: Due to the Coronavirus (COVID-19) pandemic preventing in-person data collection of task data, the N for this measure is lower than the baseline N.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Active tDCS With Cognitive Training: Participants received 5 sessions of cognitive training concurrent with transcranial direct current stimulation (anode over right frontal cortex, cathode over left frontal cortex; 2 mAmps for 26 minutes).
  Device: Active Transcranial Direct Current Stimulation (tDCS) coupled with cognitive training: Cognitive training concurrent with 2 mAmps of anodal stimulation applied to the right prefrontal cortex for total of 26 minutes.
Arm/Group | Active tDCS With Cognitive Training | Sham tDCS With Cognitive Training
Number analyzed (Participants) | 8 | 9
seconds | -0.03 (0.12) | -0.12 (0.22)

2. Primary Outcome: Change in NIH Examiner Set Shifting Task Score
Description: Difference in change in Set Shifting Task scores (score at final visit minus baseline score) between active tDCS-cognitive training and sham- Higher values represent a better outcome. Set Shifting Scale absolute value range: Minimum -10, Maximum 10.
  The Set Shifting Task Score is a combination of two subscores for reaction time and accuracy on the task.
Time Frame: Change between baseline and 4 months post-stimulation (timepoint 8, final visit)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Active tDCS With Cognitive Training: Participants will receive 5 sessions of cognitive training concurrent with transcranial direct current stimulation (anode over right frontal cortex, cathode over left frontal cortex; 2 mAmps for 26 minutes).
  Device: Active Transcranial Direct Current Stimulation (tDCS) coupled with cognitive training: Cognitive training concurrent with 2 mAmps of anodal stimulation applied to the right prefrontal cortex for total of 26 minutes.
Arm/Group | Active tDCS With Cognitive Training | Sham tDCS With Cognitive Training
Number analyzed (Participants) | 8 | 9
score on a scale | 0.46 (0.83) | 0.43 (0.74)

3. Primary Outcome: Change in NIH Examiner Dot Counting Task Score
Description: Differences in change in NIH Examiner Dot Counting Task scores (i.e., score at final visit minus baseline score) between active tDCS-cognitive training and sham-cognitive training groups. The change in score is equal to the score taken at the final follow-up visit minus the score taken at baseline.
  NIH Dot Counting absolute value range: numerical value -27 to +27. Higher values represent a better outcome.
  The Dot Count Task Score is the total sum of points awarded for dots a participant counts on the screen. The total score is a sum of scores for 27 individual trials.
Time Frame: Change between baseline and 4 months post-stimulation (i.e., timepoint 8/final visit)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS With Cognitive Training | Sham tDCS With Cognitive Training
Number analyzed (Participants) | 8 | 9
score on a scale | 2.88 (1.08) | 0.67 (1.14)

4. Primary Outcome: Change in NIH Examiner Unstructured Planning Task Score
Description: Differences in change in NIH Examiner Unstructured Planning Task scores (i.e., score at final visit minus baseline score) between active tDCS-cognitive training and sham-cognitive training groups.
  The change in score is equal to the score taken at the final follow-up visit minus the score taken at baseline. Higher values represent a better outcome.
  The Unstructured Task Score is a numeric summary score that is equal to the total sum of points awarded for completed puzzle items. The total absolute score is a sum of scores for 3 individual trials, Absolute score range :-1469 to +1469.
Time Frame: Change between baseline and 4 months post-stimulation (i.e., timepoint 8, final visit)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS With Cognitive Training | Sham tDCS With Cognitive Training
Number analyzed (Participants) | 8 | 9
score on a scale | 64.25 (41.38) | 41 (26.49)

5. Secondary Outcome: Change in Weight
Description: Difference in change in weight (pounds) between active tDCS-cognitive training and sham-cognitive training groups (i.e., end of study weight minus baseline weight).
  A more negative score indicates a better outcome.
Time Frame: Change between baseline and 4 months post-intervention (i.e., timepoint 8/final visit)
Population: Due to the Coronavirus (COVID-19) pandemic preventing in-person data collection of task data, the N for this measure is lower than the baseline N. One additional subject was excluded from the weight analysis due to participation in a commercial weight-loss program during the study.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Active tDCS With Cognitive Training | Sham tDCS With Cognitive Training
Number analyzed (Participants) | 8 | 8
pounds | 2.55 (9.33) | -6 (10.14)

6. Secondary Outcome: Effect of History of Traumatic Brain Injury on Impulsive and Compulsive Eating Behavior
Description: Effect of history of a traumatic brain injury (TBI) on impulsive/compulsive eating behavior.
  A status of either TBI+ (positive for history of TBI) or TBI- (negative for history of TBI) was determined at the baseline visit with the Minnesota Blast Exposure Screening Tool. Impulsive/compulsive eating behavior was defined as the score on the Binge Eating Scale (BES) taken at the baseline visit. Scale range = 0-48. Lower scores indicate less impulsive/compulsive eating behavior (i.e., a better outcome).
  Calculation details: Average BES scores taken at baseline for TBI-positive participants and TBI-negative participants.
Time Frame: Baseline visit
Population: Analysis was pre-specified at baseline to be reported by TBI status. Eight baseline participants did not complete the Minnesota Blast Exposure Screening Tool and were not included in this secondary analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Traumatic Brain Injury Positive (TBI+) Participants: Participants who reported having one or more traumatic brain injuries at baseline visit.
- Traumatic Brain Injury Negative (TBI-) Participants: Participants who reported having zero traumatic brain injuries at baseline visit.
Arm/Group | Traumatic Brain Injury Positive (TBI+) Participants | Traumatic Brain Injury Negative (TBI-) Participants
Number analyzed (Participants) | 6 | 17
score on a scale | 17 (8.46) | 14.94 (8.46)
Statistical Analysis 1: Comparison: Traumatic Brain Injury Positive (TBI+) Participants vs Traumatic Brain Injury Negative (TBI-) Participants; Linear regression (number of traumatic brain injuries versus Binge Eating Scale score at baseline); Test type: Other; Linear regression = 0.03

7. Post Hoc Outcome: Effect of History of Traumatic Brain Injury on Impulsive Behavior - NIH Flanker
Description: Effect of history of a traumatic brain injury (TBI) on impulsive behavior. A status of either TBI+ (positive for history of TBI) or TBI- (negative for history of TBI) was determined at baseline with the Minnesota Blast Exposure Screening Tool.
  Impulsive behavior was defined as the score on the Flanker task measured at the baseline visit. The Flanker score is equal to the average reaction time, in seconds, to respond to trials. Minimum = 0, maximum = 2. A higher score indicates less-impulsive behavior (i.e., a better outcome).
  Calculation details: Flanker scores for TBI-positive participants and TBI-negative participants.
Time Frame: Baseline visit
Population: Analysis was pre-specified at baseline to be reported by TBI status. Eight baseline participants did not complete the Minnesota Blast Exposure Screening Tool and were not included in this post-hoc analysis.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Traumatic Brain Injury-Positive (TBI+) Participants: Participants who reported having one or more Traumatic Brain Injuries at baseline visit.
- Traumatic Brain Injury-Negative (TBI-) Participants: Participants who reported having zero Traumatic Brain Injuries at baseline visit.
Arm/Group | Traumatic Brain Injury-Positive (TBI+) Participants | Traumatic Brain Injury-Negative (TBI-) Participants
Number analyzed (Participants) | 6 | 17
seconds | 0.77 (0.12) | 0.93 (0.2)
Statistical Analysis 1: Comparison: Traumatic Brain Injury-Positive (TBI+) Participants vs Traumatic Brain Injury-Negative (TBI-) Participants; Linear regression (number of traumatic brain injuries versus NIH Flanker score at baseline); Test type: Other; Linear regression = -0.33

8. Post Hoc Outcome: Effect of History of Traumatic Brain Injury on Impulsive and Compulsive Eating Behavior-NIH Set Shifting
Description: Effect of history of a traumatic brain injury (TBI) on impulsive behavior. A status of either TBI+ (positive for history of TBI) or TBI- (negative for history of TBI) was determined at baseline with the Minnesota Blast Exposure Screening Tool. Impulsive behavior was defined as the NIH Set Shifting score measured at baseline. Score range: 0 - 10. Higher scores indicate less impulsive behavior (i.e. a better outcome).
  Calculation details: Set Shifting scores for TBI-positive participants and TBI-negative participants.
Time Frame: Baseline visit
Population: Eight baseline participants did not complete the Minnesota Blast Exposure Screening Tool and were not included in this post-hoc analysis.
  Analysis was pre-specified at baseline to be reported by TBI status.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Traumatic Brain Injury Positive (TBI+) Participants | Traumatic Brain Injury Negative (TBI-) Participants
Number analyzed (Participants) | 6 | 17
score on a scale | 7.86 (0.2) | 7.75 (0.86)
Statistical Analysis 1: Comparison: Traumatic Brain Injury Positive (TBI+) Participants vs Traumatic Brain Injury Negative (TBI-) Participants; Linear regression (number of traumatic brain injuries versus NIH Set Shifting score at baseline); Test type: Other; Linear regression = 0.04

ADVERSE EVENTS:
Time Frame: Duration of treatment period (1 week)
Arm/Group | Active tDCS With Cognitive Training | Sham tDCS With Cognitive Training
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/16
Other Adverse Events (participants affected / at risk) | 10/13 | 9/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active tDCS With Cognitive Training (N=13) | Sham tDCS With Cognitive Training (N=16)
Headache (General disorders) | 4 (10) | 1 (1)
Neck pain (General disorders) | 2 (3) | 1 (1)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (1)
Tingling (General disorders) | 4 (4) | 2 (3)
Itching (General disorders) | 7 (14) | 2 (2)
Burning sensation (General disorders) | 3 (4) | 1 (1)
Skin redness (General disorders) | 6 (11) | 0 (0)
Sleepiness/fatigue (General disorders) | 5 (13) | 4 (8)
Difficulty concentrating (General disorders) | 2 (4) | 3 (7)
Acute mood change (General disorders) | 1 (1) | 2 (3)
Nausea (General disorders) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Our study was a pilot feasibility study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/89/NCT04405089/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-16): https://cdn.clinicaltrials.gov/large-docs/89/NCT04405089/ICF_002.pdf